CLINICAL TRIAL: NCT00336336
Title: A Large Scale Clinical Trial Testing the Effects of n-3 PUFA and Rosuvastatin on Mortality-Morbidity of Patients With Symptomatic Congestive Heart Failure
Brief Title: GISSI-HF- Effects of n-3 PUFA and Rosuvastatin on Mortality-Morbidity of Patients With Symptomatic CHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo di Ricerca GISSI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G105
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2010-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Fatty Acids, Omega-3; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): N-3PUFA
  Interventions: Drug: n-3 PUFA
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: n-3 PUFA — 1 g die per os
  Arms: 1
Drug: Rosuvastatin — 10 mg die per os
  Arms: 3
Drug: Placebo — 1 gram c. per os
  Arms: 2
Drug: Placebo — 10 mg c. per os
  Arms: 4

SUMMARY:
INTRODUCTION While pharmacological treatments specifically targeted to the cardio-circulatory system have been largely investigated, scanty controlled data are available concerning the role of dietary and metabolic approaches in the management/outcome of patients with heart failure. A large scale, randomized, clinical trial is proposed to test the effects of (a) n-3 PUFA and (b) a lipid lowering agent on top of the best recommended treatments for heart failure.

STUDY DESIGN

The GISSI-HF is a prospective, multicenter, randomized, double blind, placebo controlled study, with randomized allocation of patients with a clinical diagnosis of heart failure to:

Randomization 1 (R1): n-3 PUFA 1 g daily vs corresponding placebo; Randomization 2 (R2): rosuvastatin 10 mg daily vs corresponding placebo.

OBJECTIVES OF THE STUDY PRIMARY OBJECTIVES

To demonstrate that, in patients with heart failure treated at the best of recommended therapies, long term administration of (a) n-3 PUFA, (b) rosuvastatin is more effective than the corresponding placebo in the reduction of:

* All-cause mortality
* All-cause mortality or hospitalizations for cardiovascular reason

OTHER END-POINT MEASURES OF EFFICACY

To assess that long term administration of (a) n-3 PUFA, (b) rosuvastatin is more effective than corresponding placebo in the reduction of:

* Cardiovascular mortality
* Cardiovascular mortality or hospitalizations for any reason
* Sudden cardiac death
* Hospitalizations for any reason
* Hospitalizations for cardiovascular reasons
* Hospitalizations for congestive heart failure
* Myocardial infarction
* Stroke

DETAILED DESCRIPTION:
The Protocol is sponsored by an independent organization and partially supported by: AstraZeneca, Società Prodotti antibiotici, Sigma Tau, Pfizer

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of heart failure according to the European Society of Cardiology guidelines (New York Heart Association class II-IV) (32)
* Any left ventricular Ejection Fraction (EF) measured within 3 months from enrolment (if EF% >40%, at least 1 hospital admission for Congestive Heart Failure(CHF) in the previous year)
* No age limits
* Any etiology
* Informed consent (obtained before any study specific procedure)

Exclusion Criteria:

COMMON EXCLUSION CRITERIA (R1=n-3 PUFA vs placebo and R2=rosuvastatin vs placebo):

* Acute Myocardial Infarction, unstable angina or revascularization procedure within 1 month;
* planned cardiac surgery, expected to be performed within 3 months;
* congenital or primary valvular etiology;
* known hypersensitivity to study treatments;
* significant liver disease;
* pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception;
* any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety or be associated with poor adherence to the protocol;
* presence of any non-cardiac disease (e.g. cancer) that is likely to significantly shorten life expectancy;
* treatment with any investigational agent within 1 month before randomization;
* patients already on treatment with n-3 PUFA or statin for whom the prescription is confirmed.

EXCLUSION CRITERIA FOR R2 (statin hypothesis):

* current serum creatinine level >2.5 mg/dL;
* current ALT, AST level >1.5 times the upper normal limit;
* current CPK upper normal limits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6975 (Actual)
Dates: Start 2002-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | from enrollment to 1252 deaths in R2 arm
All cause mortality or hospitalizations for any reason | from enrollment to 1252 deaths

SECONDARY OUTCOMES:
Cardiovascular mortality | from enrollment to 1252 deaths in R2 arm
Cardiovascular mortality or hospitalization for heart failure or for any reasons | from enrollment to 1252 deaths in R2 arm
Sudden cardiac death | from enrollment to 1252 deaths in R2 arm
Hospitalizations for any reasons | from enrollment to 1252 deaths in R2 arm
Hospitalization for Cardiovascular reasons | from enrollment to 1252 deaths in R2 arm
Hospitalization for congestive heart failure | from enrollment to 1252 deaths in R2 arm
Miocardial infarction | from enrollment to 1252 deaths in R2 arm
Stroke | from enrollment to 1252 deaths in R2 arm

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tavazzi, MD, Study Chair — Policlinico San Matteo di Pavia; Gianni Tognoni, MD, Study Chair — Consorzio Mario Negri Sud
Locations (332):
- Italy (331):
  - Ospedale San Giovanni di Dio, Agrigento, AG
  - Ospedale Barone Lombardo, Canicattì, AG
  - Ospedale San Giacomo D'Altopasso, Licata, AG
  - Ospedale Civile, Acqui Terme, AL
  - Ospedale San Giacomo, Novi Ligure, AL
  - Presidio Cardiologico G.M. Lancisi, Ancona, AN
  - Ospedale Generale Regionale, Aosta, AO
  - Osp. Gen.le Prov.le C.G.Mazzoni, Ascoli Piceno, AP
  - Ospedale Civile Augusto Murri, Fermo, AP
  - Ospedale Madonna del Soccorso, San Benedetto del Tronto, AP
  - Ospedale Civile SS.Filippo e Nicola, Avezzano, AQ
  - Presidio Ospedaliero San Salvatore, L’Aquila, AQ
  - Ospedale San Donato, Arezzo, AR
  - Ospedale Valdichiana Santa Margherita, Cortona, AR
  - Osp.Valdarno "S.Maria della Gruccia", Montevarchi, AR
  - Ospedale Cardinal Massaia, Asti, AT
  - Ospedale San Paolo, Bari, BA
  - Ospedale Consorziale Policlinico, Bari, BA
  - Ospedale di Venere, Bari - Carbonara, BA
  - Ospedale Monsignor Angelo R. di Miccoli, Barletta, BA
  - Fondazione S. Maugeri Clinica del Lavoro, Cassano delle Murge, BA
  - IRCCS Saverio De Bellis, Castellana Grotte, BA
  - Ospedale Santa Maria degli Angeli, Putignano, BA
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Ospedale Bolognini, Seriate, BG
  - Presidio Gazzaniga c/o Osp. Seriate, Seriate, BG
  - Ospedali Riuniti di Treviglio, Treviglio, BG
  - Ospedale Civile, Agordo, BL
  - Ospedale Civile, Belluno, BL
  - Ospedale Civile del Cadore, Pieve di Cadore, BL
  - Ospedale Dossetti, Bazzano, BO
  - Ospedale di Bentivoglio, Bentivoglio, BO
  - Ospedale Policlinico S.Orsola-M.Malpighi, Bologna, BO
  - Ospedale Bellaria, Bologna, BO
  - Ospedale Civile Simiani, Loiano, BO
  - Ospedale Umberto I, Fasano, BR
  - Ospedale Civile Dario Camberlingo, Francavilla Fontana, BR
  - Ospedale N. Melli, San Pietro Vernotico, BR
  - Spedali Civili, Brescia, BS
  - Ospedale Civile Mellini, Chiari, BS
  - Azienda Ospedaliera, Desenzano del Garda, BS
  - Presidio Ospedaliero, Gavardo, BS
  - Ospedale di Manerbio, Manerbio, BS
  - Ospedale Generale Provinciale, Merano, BZ
  - Osedale A. Businco, Cagliari, CA
  - Presidio Ospedaliero SS. Trinita', Cagliari, CA
  - Ospedale Marino, Cagliari, CA
  - Azienda Osped. G.Brotzu-S.Michele (S.S.D.coord.Scompenso), Cagliari, CA
  - Azienda Ospedaliera G. Brotzu - S. Michele, Cagliari, CA
  - Universita', Cagliari-Monserrato, CA
  - Ospedale Civile G. Vietri, Larino, CB
  - Ospedale San Timoteo, Termoli, CB
  - Presidio Ospedaliero Moscati, Aversa, CE
  - Az. Ospedaliera S.Anna e S.Sebastiano, Caserta, CE
  - Azienda Ospedaliera Sant'Anna e San Sebastiano, Caserta, CE
  - P.O. Marcianese ASL Caserta 1, Marcianise, CE
  - Ospedale Civile Ave Gratia Plena, Piedimonte Matese, CE
  - Ospedale Ave Gratia Plena, San Felice A Cancello, CE
  - Ospedale Renzetti, Lanciano, CH
  - Ospedale San Pio da Pietrelcina, Vasto, CH
  - Ospedale Civile San Lazzaro, Alba, CN
  - Ospedale Maggiore SS. Trinita', Fossano, CN
  - Ospedale Civile Saluzzo, Saluzzo, CN
  - Ospedale Generale di Zona Valduce, Como, CO
  - Ospedale S. Anna, Como, CO
  - A.O. S. Anna-Presidio di Mariano Comense, Mariano Comense, Co
  - Ospedale di Menaggio, Menaggio, CO
  - Ospedale Civile Oglio Po, Casalmaggiore, CR
  - Istituti Ospitalieri di Cremona, Cremona, CR
  - Ospedale Santa Marta, Rivolta d'Adda, CR
  - Ospedale V. Cosentino, Cariati, CS
  - Ospedale Civile Ferrari, Castrovillari, CS
  - Ospedale Civile Guido Compagna, Corigliano Calabro, CS
  - INRCA Istituto Cardiovasculop.Senili, Cosenza, CS
  - Ospedale Santissima Annunziata, Cosenza, CS
  - Presidio Ospedaliero Mariano Santo, Cosenza, CS
  - Ospedale Civile Minervini, Mormanno, CS
  - Ospedale San Francesco di Paola, Paola, CS
  - Ospedale Santa Barbara, Rogliano, CS
  - Ospedale Civile N. Giannettasio, Rossano, CS
  - Ospedale Civile G. Chidichimo, Trebisacce, CS
  - Ospedale Generale Provinciale Gravina, Caltagirone, CT
  - Ospedale Garibaldi - Nesima, Catania, CT
  - Ospedale Garibaldi-Nesima, Catania, CT
  - Ospedale Ferrarotto, Catania, CT
  - Ospedale Garibaldi - Centro, Catania, CT
  - Ospedale Vittorio Emanuele II, Catania, CT
  - Ospedale Cannizzaro (U.O.Cardiologia), Catania, CT
  - Ospedle Cannizzaro (UTIC), Catania, CT
  - Azienda Ospedaliera Mater Domini, Catanzaro, CZ
  - Ospedale Civile Pugliese, Catanzaro, CZ
  - Azienda Ospedaliera Mater Domini, Località Germaneto - Catanzaro, CZ
  - Ospedale G. Basilotta, Nicosia, EN
  - Ospedale M. Chiello, Piazza Armerina, EN
  - Ospedale M. Bufalini-G. Marconi, Cesena, FC
  - Ospedale M.Bufalini-G.Marconi, Cesenatico, FC
  - Ospedale G.B.Morgagni-L.Pierantoni, Forlì, FC
  - Arcispedale Sant'Anna, Ferrara, FE
  - Ospedale del Delta, Lagosanto, FE
  - Ospedale Civile Giuseppe Tatarella, Cerignola, FG
  - Ospedali Riuniti, Foggia, FG
  - Ospedale San Camillo De Lellis, Manfredonia, FG
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, FI
  - Presidio Ospedaliero del Mugello, Borgo San Lorenzo, FI
  - Ospedale Civile San Giuseppe, Empoli, FI
  - Ospedale Santa Maria Nuova, Florence, FI
  - Presidio Ospedaliero di Camerata, Florence, FI
  - Az. Ospedaliero-Universitaria Careggi, Florence, FI
  - Nuovo Ospedale San Giovanni di Dio, Florence, FI
  - Ospedale San Pietro Igneo, Fucecchio, FI
  - Ospedale Santa Scolastica, Cassino, FR
  - Ospedale Civile SS. Trinita', Sora, FR
  - Dimi-Disem, Genova, GE
  - Ospedali Civili di Sampierdarena, Genova-Sampierdarena, GE
  - Ospedale Padre Antero Micone, Genova-Sestri Ponente, GE
  - Ospedale Sestri Levante, Sestri Levante, GE
  - Presidio Ospedaliero di Gorizia, Gorizia, GO
  - Ospedale della Misericordia, Grosseto, GR
  - Ospedale S.Andrea-Alta Maremma, Massa Marittima, GR
  - Ospedale San Giovanni di Dio, Orbetello, GR
  - Presidio Ospedaliero, Sanremo, IM
  - Ospedale F. Veneziale, Isernia, IS
  - Ospedale Civile San Giovanni di Dio, Crotone, KR
  - Ospedale di Mesoraca, Mesoraca, KR
  - Ospedale Umberto I, Lecco, LC
  - Presidio Ospedaliero F. Ferrari, Casarano, LE
  - Ospedale Santa Caterina Novella, Galatina, LE
  - Ospedale Civile Sacro Cuore di Gesu', Gallipoli, LE
  - Ospedale Vito Fazzi, Lecce, LE
  - Presidio Osped. Pneumologico Galateo, San Cesario di Lecce, LE
  - Ospedale Ignazio Veris Delli Ponti, Scorrano, LE
  - Ospedale Cardinale Panico, Tricase, LE
  - Ospedale Civile Bassa Val di Cecina, Cecina, LI
  - Ospedali Riuniti, Livorno, LI
  - Ospedale Villamarina, Piombino, LI
  - Ospedale del dono Svizzero, Formia, LT
  - Ospedale Civile, Gaeta, LT
  - Ospedale S. Maria Goretti, Latina, LT
  - Ospedale Generale di Zona, Minturno, LT
  - Ospedale Civile, Terracina, LT
  - Ospedale Santa Croce, Castelnuovo Garfagnana, LU
  - Nuovo Ospedale Versilia, Lido di Camaiore, LU
  - Ospedale Santa Maria della Pieta', Camerino, MC
  - Ospedale Generale Provinciale, Macerata, MC
  - Nuovo Pres.Osp. Cutroni Zodda, Barcellona Pozzo di Gotto, ME
  - Ospedale Papardo, Messina, ME
  - Ospedale Civile, Milazzo, ME
  - Ospedale Barone Romeo, Patti, ME
  - P.O. Sant'Agata di Militello, Sant'Agata di Militello, ME
  - Presidio Ospedaliero San Vincenzo, Taormina, ME
  - Ospedale di Cernusco sul Naviglio, Cernusco sul Naviglio, MI
  - Ospedale Carlo Borella, Giussano, MI
  - Ospedale Civile, Legnano, MI
  - Ospedale Fatebenefratelli, Milan, MI
  - Ospedale Maggiore Policlinico, Milan, MI
  - Centro Cardiologico Monzino, Milan, MI
  - Ospedale San Paolo, Milan, MI
  - Ospedale San Carlo Borromeo, Milan, MI
  - Ospedale Niguarda-Villa Marelli, Milan, MI
  - Ospedale Niguarda, Milan, MI
  - Ospedale San Gerardo, Monza, MI
  - Policlinico di Monza, Monza, MI
  - Presidio Ospedaliero di Passirana, Passirana-Rho, MI
  - Ospedale di Sesto San Giovanni, Sesto San Giovanni, MI
  - Presidio Ospedaliero, Vimercate, MI
  - Ospedale di Vizzolo Predabissi, Vizzolo Predabissi, MI
  - Ospedale San Pellegrino, Castiglione delle Stiviere, MN
  - Presidio Ospedaliero C. Poma, Mantova, MN
  - Ospedali Destra Secchia, Pieve di Coriano, MN
  - Ospedale Policlinico, Modena, MO
  - Presidio Ospedaliero, Pavullo nel Frignano, MO
  - Nuovo Ospedale Civile di Sassuolo, Sassuolo, MO
  - Civico Ospedale Carrara, Carrara, MS
  - IFC CNR-Ospedale Pasquinucci, Massa, MS
  - Ospedale SS.Giacomo e Cristoforo, Massa, MS
  - Ospedale Madonna delle Grazie, Matera, MT
  - Ospedale Civile, Policoro, MT
  - Ospedale San Francesco, Nuoro, NU
  - Fondazione San Raffaele G. Giglio, Cefalù, PA
  - Ospedale Buccheri La Ferla Fatebenefratelli, Palermo, PA
  - A.R.N.A.S. Ospedale Civico e Benfratelli, Palermo, PA
  - Ospedale G.F. Ingrassia, Palermo, PA
  - Az. Osp. Villa Sofia CTO (Cardiologia II), Palermo, PA
  - Ospedale V. Cervello, Palermo, PA
  - Presidio Ospedaliero Villa Sofia, Palermo, PA
  - Ospedale Pubblico S. Cimino, Termini Imerese, PA
  - Ospedale di Camposampiero, Camposampiero, PD
  - Ospedale di Cittadella, Cittadella, PD
  - Ospedale Generale Provinciale, Este, PD
  - Ospedale Civile San Massimo, Penne, PE
  - Ospedale Civile dello Spirito Santo, Pescara, PE
  - Ospedale Alta Valle del Tevere, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista, Foligno, PG
  - Ospedale Gubbio-Gualdo Tadino, Gubbio, PG
  - Centro Osp.Riabilit.Intensiva (CORI), Passignano sul Trasimeno, PG
  - Presidio Ospedaliero, Todi, PG
  - Azienda Ospedaliera S. Maria degli Angeli, Pordenone, PN
  - Ospedale Civile, San Vito al Tagliamento, PN
  - Ospedale Misericordia e Dolce, Prato, PO
  - Ospedale Civile, Fidenza, PR
  - Az. Ospedaliera Universitaria di Parma, Parma, PR
  - Ospedale Santa Maria della Misericordia, Urbino, PU
  - Ospedale San Martino, Mede, PV
  - Fondazione S.Maugeri Clinica del Lavoro, Montescano, PV
  - IRCCS - Fondazione Salvatore Maugeri, Pavia, PV
  - Ospedale Policlinico San Matteo IRCCS, Pavia, PV
  - Istituto Clinico Beato Matteo, Vigevano, PV
  - Ospedale Civile, Vigevano, PV
  - Ospedale Civile, Voghera, PV
  - Ospedale Generale di Zona, Lagonegro, PZ
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Ospedale San Francesco, Venosa, PZ
  - Villa Maria Cecilia Hospital, Cotignola, RA
  - Policlinico Madonna della Consolazione, Reggio Calabria, RC
  - Ospedale Scillesi D'America, Scilla, RC
  - Ospedale Sant'Anna, Castelnovo ne' Monti, Re
  - Ospedale Civile San Sebastiano, Correggio, RE
  - Ospedale Civile, Ragusa, RG
  - Ospedale M.P. Arezzo, Ragusa, RG
  - P.O. San Camillo De Lellis, Rieti, RI
  - Ospedali Riuniti Albano-Genzano, Albano Laziale, RM
  - Ospedale Civile San Paolo, Civitavecchia, RM
  - Ospedale Generale Zona Parodi Delfino, Colleferro, RM
  - Ospedale San Sebastiano Martire, Frascati, RM
  - Ospedale San Giuseppe, Marino, RM
  - Ospedale di Monterotondo, Monterotondo, RM
  - Campus Biomedico, Roma, RM
  - Ospedale San Filippo Neri, Roma, RM
  - Ospedale Sant'Eugenio, Roma, RM
  - Ospedale C. Forlanini, Roma, RM
  - Ospedale San Camillo, Roma, RM
  - Ospedale Sandro Pertini, Roma, RM
  - Policlinico Umberto Primo, Roma, RM
  - Ospedale San Carlo di Nancy, Roma, RM
  - Presidio Ospedaliero Villa Betania, Roma, RM
  - Ospedale Generale di Zona "Cristo Re", Roma, RM
  - Ospedale Fatebenefratelli, Roma, RM
  - Policlinico Agostino Gemelli, Roma, RM
  - I.N.R.C.A., Roma, RM
  - Ospedale Santo Spirito, Roma, RM
  - Ospedale A. Angelucci, Subiaco, RM
  - Ospedale San Giovanni Evangelista, Tivoli, RM
  - Ospedale Civile, Velletri, RM
  - Ospedale G. Ceccarini, Riccione, RN
  - Ospedale Infermi, Rimini, RN
  - Ospedale Civile, Adria, RO
  - Presidio Ospedaliero, Rovigo, RO
  - Presidio Ospedaliero S.Maria della Speranza, Battipaglia, SA
  - Ospedale G. Fucito, Mercato San Severino, SA
  - Ospedale Civile, Nocera Inferiore, SA
  - Ospedale San Francesco D'Assisi, Oliveto Citra, SA
  - A.O. S.Giovanni di Dio e Ruggi di Aragona, Salerno, SA
  - Ospedale dell'Immacolata, Sapri, SA
  - Ospedale Civile, Scafati, SA
  - Ospedale San Luca, Vallo della Lucania, SA
  - Presidio Ospedaliero Valdichiana Senese, Montepulciano, SI
  - Presidio Ospedaliero, Poggibonsi, SI
  - Policlinico Santa Maria alle Scotte, Siena, SI
  - Ospedale Civile, Morbegno, SO
  - Ospedale E. Morelli, Sondalo, SO
  - Ospedale Civile, Sondrio, SO
  - Ospedale S. Andrea, La Spezia, SP
  - Ospedale San Bartolomeo, Sarzana - Loc. Santa Caterina, SP
  - Azienda Ospedaliera Umberto I, Syracuse, SR
  - Az. Ospedaliero Universitaria di Sassari, Sassari, SS
  - Ospedale Civile, Thiesi, SS
  - Ospedale Civile, Castellaneta, TA
  - Presidio Ospedaliero della Valle D'Itria, Martina Franca, TA
  - Ospedale Umberto I, Mottola, TA
  - Ospedale S. Giuseppe Moscati, Taranto, TA
  - Ospedale SS. Annunziata, Taranto, TA
  - Ospedale Civile G. Mazzini, Teramo, TE
  - Ospedale Alto Garda e Ledro, Arco, TN
  - Casa di Cura Villa Bianca, Trento, TN
  - Ospedale Santa Croce, Moncalieri, To
  - Ospedale San Luigi Gonzaga, Orbassano, TO
  - Ospedale Civile E. Agnelli, Pinerolo, TO
  - Presidio Ospedaliero, Susa, TO
  - Ospedale Evangelico Valdese, Torino, TO
  - Ospedale Martini, Torino, TO
  - Ospedale Maria Vittoria, Torino, TO
  - Presidio Ospedaliero Gradenigo, Torino, TO
  - Ospedale Civile Vittorio Emanuele II, Castelvetrano, TP
  - Ospedale Civile Sant'Antonio Abate, Erice, TP
  - Ospedale A. Ajello, Mazara del Vallo, TP
  - Azienda USL 4 Terni, Terni, TR
  - Azienda Ospedaliera - Univ. Ospedali Riuniti, Trieste, TS
  - Ospedale De Gironcoli, Conegliano Veneto, TV
  - Ospedale Santa Maria dei Battuti, Conegliano Veneto, TV
  - Ospedale Ca' Foncello, Treviso, TV
  - Ospedale di Ialmicco - Palmanova - Udine, Palmanova, UD
  - Ospedale S. Antonio, San Daniele del Friuli, UD
  - Ospedale Civile Sant'Antonio Abate, Tolmezzo, UD
  - Santa Maria della Misericordia, Udine, UD
  - Ospedale S. Antonio Abate, Gallarate, VA
  - Presidio Ospedaliero, Saronno, VA
  - Ospedale di Circolo A. Bellini, Somma Lombardo, VA
  - Fondazione S. Maugeri Clinica del Lavoro, Tradate, VA
  - Azienda Ospedaliera e Universitaria, Varese, VA
  - Ospedale del Ponte, Varese, VA
  - Ospedale Castelli, Verbania, VB
  - Ospedale Civile, Dolo, VE
  - Ospedale Civile Umberto I, Mestre, VE
  - Ospedale Civile, Mirano, VE
  - Ospedale Civile, Portogruaro, VE
  - Ospedali Civili Riuniti, Venezia, VE
  - Ospedale Civile, Noventa Vicentina, VI
  - Ospedale Civile San Biagio, Bovolone, VR
  - Ospedale Mater Salutis, Legnago, VR
  - Ospedale Sacro Cuore, Negrar, VR
  - Ospedale G. Fra Castoro, San Bonifacio, VR
  - Azienda Ospedaliera, Verona, VR
  - Ospedale di Villafranca, Villafranca di Verona, VR
  - Presidio Ospedaliero, Soriano Calabro, VV
  - Ospedale Civile G. Jazzolino, Vibo Valentia, VV
  - Ospedale SS. Trinita', Borgomanero
  - Ospedale Civile di Boscotrecase, Boscotrecase
  - Opsedale San Leonardo, Castellammare di Stabia
  - Ospedale Civile San Giovanni di Dio, Frattaminore
  - Ospedale Generale di Zona, Giugliano in Campania
  - MIOspedale San Raffaele, Milan
  - AORN Cardarelli, Napoli
  - Azienda Ospedaliera Vincenzo Monaldi, Napoli
  - Fondazione Pascale, Napoli
  - Ospedale Domenico Cotugno, Napoli
  - Policlinico Universitario Federico II, Napoli
  - Pres.Ospedaliero S. Maria della Pieta', Nola
  - Ospedale Santa Maria delle Grazie, Pozzuoli
  - Ospedale Santa Maria della Misericordia, Sorrento
  - Fondazione Salvatore Maugeri, Veruno
- Cardiocentro Ticino, Lugano, Switzerland

REFERENCES:
- [Background] Tavazzi L, Tognoni G, Franzosi MG, Latini R, Maggioni AP, Marchioli R, Nicolosi GL, Porcu M; GISSI-HF Investigators. Rationale and design of the GISSI heart failure trial: a large trial to assess the effects of n-3 polyunsaturated fatty acids and rosuvastatin in symptomatic congestive heart failure. Eur J Heart Fail. 2004 Aug;6(5):635-41. doi: 10.1016/j.ejheart.2004.03.001. PMID 15302013
- [Result] Tavazzi L, Maggioni AP, Marchioli R, Barlera S, Franzosi MG, Latini R, Lucci D, Nicolosi GL, Porcu M, Tognoni G; Gissi-HF Investigators. Effect of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Oct 4;372(9645):1223-30. doi: 10.1016/S0140-6736(08)61239-8. Epub 2008 Aug 29. PMID 18757090
- [Result] Tavazzi L, Maggioni AP, Marchioli R, Barlera S, Franzosi MG, Latini R, Lucci D, Nicolosi GL, Porcu M, Tognoni G; Gissi-HF Investigators. Effect of rosuvastatin in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Oct 4;372(9645):1231-9. doi: 10.1016/S0140-6736(08)61240-4. Epub 2008 Aug 29. PMID 18757089
- [Derived] Canepa M, Ameri P, Lucci D, Nicolosi GL, Marchioli R, Porcu M, Tognoni G, Franzosi MG, Latini R, Maseri A, Tavazzi L, Maggioni AP; GISSI-HF Investigators. Modes of death and prognostic outliers in chronic heart failure. Am Heart J. 2019 Feb;208:100-109. doi: 10.1016/j.ahj.2018.11.009. Epub 2018 Nov 24. PMID 30580128
- [Derived] Mantovani A, Targher G, Temporelli PL, Lucci D, Gonzini L, Nicolosi GL, Marchioli R, Tognoni G, Latini R, Cosmi F, Tavazzi L, Maggioni AP; GISSI-HF Investigators. Prognostic impact of elevated serum uric acid levels on long-term outcomes in patients with chronic heart failure: A post-hoc analysis of the GISSI-HF (Gruppo Italiano per lo Studio della Sopravvivenza nella Insufficienza Cardiaca-Heart Failure) trial. Metabolism. 2018 Jun;83:205-215. doi: 10.1016/j.metabol.2018.02.007. Epub 2018 Mar 29. PMID 29477817
- [Derived] Dauriz M, Targher G, Temporelli PL, Lucci D, Gonzini L, Nicolosi GL, Marchioli R, Tognoni G, Latini R, Cosmi F, Tavazzi L, Maggioni AP; GISSI-HF Investigators. Prognostic Impact of Diabetes and Prediabetes on Survival Outcomes in Patients With Chronic Heart Failure: A Post-Hoc Analysis of the GISSI-HF (Gruppo Italiano per lo Studio della Sopravvivenza nella Insufficienza Cardiaca-Heart Failure) Trial. J Am Heart Assoc. 2017 Jul 5;6(7):e005156. doi: 10.1161/JAHA.116.005156. PMID 28679559
- [Derived] Rossi A, Inciardi RM, Rossi A, Temporelli PL, Lucci D, Gonzini L, Marchioli R, Nicolosi GL, Tavazzi L; GISSI-HF Investigators. Prognostic effects of rosuvastatin in patients with co-existing chronic obstructive pulmonary disease and chronic heart failure: A sub-analysis of GISSI-HF trial. Pulm Pharmacol Ther. 2017 Jun;44:16-23. doi: 10.1016/j.pupt.2017.03.001. Epub 2017 Mar 3. PMID 28263812
- [Derived] Florea VG, Rector TS, Anand IS, Cohn JN. Heart Failure With Improved Ejection Fraction: Clinical Characteristics, Correlates of Recovery, and Survival: Results From the Valsartan Heart Failure Trial. Circ Heart Fail. 2016 Jul;9(7):e003123. doi: 10.1161/CIRCHEARTFAILURE.116.003123. PMID 27413037
- [Derived] Damman K, Masson S, Hillege HL, Voors AA, van Veldhuisen DJ, Rossignol P, Proietti G, Barbuzzi S, Nicolosi GL, Tavazzi L, Maggioni AP, Latini R. Tubular damage and worsening renal function in chronic heart failure. JACC Heart Fail. 2013 Oct;1(5):417-24. doi: 10.1016/j.jchf.2013.05.007. Epub 2013 Sep 11. PMID 24621973
- [Derived] Barlera S, Tavazzi L, Franzosi MG, Marchioli R, Raimondi E, Masson S, Urso R, Lucci D, Nicolosi GL, Maggioni AP, Tognoni G; GISSI-HF Investigators. Predictors of mortality in 6975 patients with chronic heart failure in the Gruppo Italiano per lo Studio della Streptochinasi nell'Infarto Miocardico-Heart Failure trial: proposal for a nomogram. Circ Heart Fail. 2013 Jan;6(1):31-9. doi: 10.1161/CIRCHEARTFAILURE.112.967828. Epub 2012 Nov 14. PMID 23152490
- [Derived] La Rovere MT, Pinna GD, Maestri R, Barlera S, Bernardinangeli M, Veniani M, Nicolosi GL, Marchioli R, Tavazzi L; GISSI-HF Investigators. Autonomic markers and cardiovascular and arrhythmic events in heart failure patients: still a place in prognostication? Data from the GISSI-HF trial. Eur J Heart Fail. 2012 Dec;14(12):1410-9. doi: 10.1093/eurjhf/hfs126. Epub 2012 Jul 30. PMID 22851700
- [Derived] Latini R, Gullestad L, Masson S, Nymo SH, Ueland T, Cuccovillo I, Vardal M, Bottazzi B, Mantovani A, Lucci D, Masuda N, Sudo Y, Wikstrand J, Tognoni G, Aukrust P, Tavazzi L; Investigators of the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA) and GISSI-Heart Failure (GISSI-HF) trials. Pentraxin-3 in chronic heart failure: the CORONA and GISSI-HF trials. Eur J Heart Fail. 2012 Sep;14(9):992-9. doi: 10.1093/eurjhf/hfs092. Epub 2012 Jun 27. PMID 22740508
- [Derived] Masson S, Anand I, Favero C, Barlera S, Vago T, Bertocchi F, Maggioni AP, Tavazzi L, Tognoni G, Cohn JN, Latini R; Valsartan Heart Failure Trial (Val-HeFT) and Gruppo Italiano per lo Studio della Sopravvivenza nell'Insufficienza Cardiaca-Heart Failure (GISSI-HF) Investigators. Serial measurement of cardiac troponin T using a highly sensitive assay in patients with chronic heart failure: data from 2 large randomized clinical trials. Circulation. 2012 Jan 17;125(2):280-8. doi: 10.1161/CIRCULATIONAHA.111.044149. Epub 2011 Dec 2. PMID 22139751
- [Derived] Damman K, Masson S, Hillege HL, Maggioni AP, Voors AA, Opasich C, van Veldhuisen DJ, Montagna L, Cosmi F, Tognoni G, Tavazzi L, Latini R. Clinical outcome of renal tubular damage in chronic heart failure. Eur Heart J. 2011 Nov;32(21):2705-12. doi: 10.1093/eurheartj/ehr190. Epub 2011 Jun 11. PMID 21666249
- [Derived] Finzi AA, Latini R, Barlera S, Rossi MG, Ruggeri A, Mezzani A, Favero C, Franzosi MG, Serra D, Lucci D, Bianchini F, Bernasconi R, Maggioni AP, Nicolosi G, Porcu M, Tognoni G, Tavazzi L, Marchioli R. Effects of n-3 polyunsaturated fatty acids on malignant ventricular arrhythmias in patients with chronic heart failure and implantable cardioverter-defibrillators: A substudy of the Gruppo Italiano per lo Studio della Sopravvivenza nell'Insufficienza Cardiaca (GISSI-HF) trial. Am Heart J. 2011 Feb;161(2):338-343.e1. doi: 10.1016/j.ahj.2010.10.032. PMID 21315217
- [Derived] Maggioni AP, Fabbri G, Lucci D, Marchioli R, Franzosi MG, Latini R, Nicolosi GL, Porcu M, Cosmi F, Stefanelli S, Tognoni G, Tavazzi L; GISSI-HF Investigators. Effects of rosuvastatin on atrial fibrillation occurrence: ancillary results of the GISSI-HF trial. Eur Heart J. 2009 Oct;30(19):2327-36. doi: 10.1093/eurheartj/ehp357. Epub 2009 Aug 30. PMID 19717850
- See also: Related Info — http://www.gissi.org
- See also: Related Info — http://www.anmco.it